CLINICAL TRIAL: NCT00989300
Title: Influence of Rabeprazole on the Magnitude of the Antiplatelet Action of Clopidogrel. A Prospective, placebo-and Active Treatment-controlled, Open Label, Randomized 3-way Cross Over Study in Healthy Subjects
Brief Title: Influence of Rabeprazole on the Magnitude of the Antiplatelet Action of Clopidogrel
Acronym: CLARA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Cilag S.A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR016333; RABGRD1008 (Other: Janssen-Cilag International NV); 2009-014756-29 (EudraCT Number)
Record Dates: First submitted 2009-10-02; First posted 2009-10-05 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Drug-Drug interaction; Clopidogrel; Rabeprazol; Omeprazol; Pharmacodynamic Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group (Experimental): patients received clopidogrel 75 mg with rabeprazole 20 mg, omeprazole 20 mg, or placebo in a crossover manner
  Interventions: Drug: Treatment A - rabeprazole; Drug: Treatment B - omeprazole
- Placebo group (Placebo Comparator)
  Interventions: Other: Treatment C - placebo

INTERVENTIONS:
Drug: Treatment A - rabeprazole — 20 mg rabeprazole sodium once daily for 7 days, in combination with 75 mg clopidogrel once daily for 7 days, oral dosing
  Arms: Treatment group
Drug: Treatment B - omeprazole — 20 mg omeprazole once daily for 7 days, in combination with 75 mg clopidogrel once daily for 7 days, oral dosing
  Arms: Treatment group
Other: Treatment C - placebo — placebo once daily for 7 days, in combination with 75 mg clopidogrel once daily for 7 days, oral dosing
  Arms: Placebo group

SUMMARY:
The purpose of this study is to assess, whether the administration of a proton pump inhibitor, Rabeprazole, has a negative effect on the activity of a concomitantly administered blood thinner drug. Proton pump inhibitors (PPI's) are prescribed for patients with gastric problems to reduce the gastric acid secretion. The blood thinner drug, Clopidogrel, administered in this trial is approved for the treatment of mild heart attacks; it works by preventing blood platelets from sticking together to form clots that would restrict blood flow. Previous trials have shown that the proton pump inhibitor omeprazole interacts with the blood thinning drug clopidogrel to reduce the active form of clopidogrel, thereby preventing the drug's blood thinning effect. In this trial, the effect of two different proton pump inhibitors, namely rabeprazole and omeprazole on the activity of the blood thinner drug clopidogrel will be assessed and compared to the effect of placebo on the activity of the blood thinner drug clopidogrel. This will be done in three sequential periods and each of the patients enrolled into this trial will be asked to participate in three different periods, during which clopidogrel with either rabeprazol, or omeprazol, or placebo will be administered daily.

DETAILED DESCRIPTION:
In this open-label trial (investigators and patients know, what medication is administered), participants will in the course of three different periods, receive three different combinations of study drugs, namely either clopidogrel combined with rabeprazole, or clopidogrel combined with omeprazole or clopidogrel combined with placebo. Each of these treatment periods will last 7 days and will be interrupted by 2 to 3 weeks without any medication. The goal is to recruit a total of 36 healthy volunteers for all three periods. Clopidogrel is a blood thinner drug that acts on the platelet cell membrane. By this mechanism, clopidogrel inhibits the platelets aggregation. Clopidogrel is a prodrug, meaning that it is orally administrated as an inactive drug and must be activated through several biochemical steps to acquire its antiplatelet properties. This process takes place in the liver and implies a complex enzymatic system. A part of this enzymatic system, called cytochrome 2C19 (CYP2C19) has an important role in the metabolism of the clopidogrel and of other drugs. One of the drugs, which is also metabolized through this system is the proton pump inhibitor (PPI) omeprazole. If omeprazole is given concomitantly with clopidogrel, the metabolism of clopidogrel is inhibited and as a consequence, the therapeutic activity of clopidogrel is reduced. The aim of this study is to investigate whether the proton pump inhibitor rabeprazole, whose metabolism is much less dependent on CYP2C19, interferes less with clopidogrel bioactivation and could thus be proposed as an alternative to other PPIs to patients taking clopidogrel. To confirm that rabeprazole has no clinically relevant effect on the metabolism of clopidogrel, one session is performed with placebo tablets in combination with clopidogrel. Each patient will receive 2 types of study drug during 3 separate periods; either one tablet clopidogrel (75 mg) combined with rabeprazole, or clopidogrel (75 mg) combined with omeprazole or clopidogrel (75 mg) combined with placebo. Each of these treatment periods will last 7 days and will be interrupted by 2 to 3 weeks without any medication.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer in good health as determined by a medical history, physical examination including vital signs, and clinical laboratory test results
* Body Mass Index between 18 and 30 kg/m2 (inclusive) and body weight not less than 50 kg
* Non smoker or smokes <5 cigarettes /day, at least 6 months before first study drug
* ECG, blood pressure in normal range (blood pressure measured after the subject is sitting for 5 minutes, between 90 and 140 mm Hg systolic (inclusive) and no higher than 90 mmHg diastolic)

Exclusion Criteria:

* Personal or family history of coagulation or bleeding disorders
* Use of known inhibitors or inducers of CYP2C19 and CYP3A, including grape fruit juice intake
* Use of any prescription or non prescription medication (including vitamins and herbal supplements), except for paracetamol (acetaminophen) within 14 days prior to screening
* Known hypersensitivity to clopidogrel, rabeprazole, its excipients, omeprazole or substituted benzimidazoles
* Current clinically significant medical illness or history of clinically significant medical illness
* History of, or reason to believe a volunteer has a history of drug or alcohol abuse within the past 5 years

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-11; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The effect of rabeprazole and placebo on inhibition of platelet function after 7 daily standard 75 mg doses of clopidogrel in healthy male volunteers. | Day 7 of period 1, 2 or 3

SECONDARY OUTCOMES:
The difference in inhibiting the activity of clopidogrel after the administration of rabeprazole compared to placebo | Measurement at day 7 of period 1, 2 or 3
The difference in inhibiting the activity of clopidogrel after the administration of omeprazole compared to placebo | measurement at day 7 of period 1, 2, or 3
The difference in inhibiting the activity of clopidogrel after the administration of rabeprazole compared to omeprazole. | measurement at day 7 of period 1, 2, or 3

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.A.S. Clinical Trial, Study Director — Janssen Cilag S.A.S.

REFERENCES:
- See also: Influence of rabeprazole on the magnitude of the antiplatelet action of clopidogrel. A prospective, placebo and active treatment-controlled, open-label, randomized 3-way cross over study in healthy subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=275&filename=CR016333_CSR.pdf